CLINICAL TRIAL: NCT01307540
Title: Phototherapy for the Management of Oral Ulcers in Bone Marrow Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Sharon Elad, PI, Hadassah University Medical Center
Allocation: Randomized | Masking: Triple | Purpose: Prevention
Other Study IDs: HT3687
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2010-06

CONDITIONS: Oral Mucosal Ulceration; Oral Mucositis; Oral Lesion
MeSH Terms: conditions — Oral Ulcer; Stomatitis | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Active light therapy (Experimental): oral mucosa is exposed to a light source (broad band of wavelengths, 400-800 nm)
  Interventions: Device: phototherapy
- Inactive light therapy (Placebo Comparator): Oral mucosa is exposed to a extremely low-intensity light which is assumed to have no effect.
  Interventions: Device: phototherapy

INTERVENTIONS:
Device: phototherapy — low level light therapy, broad band light wavelengths.
  Other Names: QRay1

SUMMARY:
Study hypothesis: light therapy may prevent oral ulcers in bone marrow recipients.

Methods: patients will be treated with either active light-emitting device or inactive light-emitting device. Daily treatment with light therapy will start at the beginning of the conditioning regimen and will last until day 21 post-transplant. Each daily treatment last about 5 minutes. Patients will be evaluated for oral mucositis and oral pain level on a weekly basis.

DETAILED DESCRIPTION:
Primary endpoint:

o Assessment of effectiveness of treatment with QRay1 in preventing oral mucositis in patients undergoing hematopoietic stem cell transplantation (HSCT).

Secondary endpoint:

* Assessment of mucositis associated- pain relief.
* Assessment of safety of treatment with QRay1 (oral adverse events).
* Assessment of the patients' acceptance of the device.

Study design:

Double-blind, randomized, placebo-controlled, 2 groups (randomization ratio 1:1).

Duration of treatment:

Daily treatment. Study-treatment administration began at the initiation of conditioning regimen (visit 1) and continued to day 28 or at least until day 21 if the patient had no mucositis (WHO or OMAS = "0")

Light radiation dose:

60-70mW/cm2 (administered over 3 treatment areas), starting with 45 seconds per surface, increasing each day in intervals of 15 seconds, up to a maximum of 90 seconds per surface.

Evaluation plan:

Evaluation began before the conditioning regimen was initiated (visit 1) and continued weekly until day 28 or until day 21 if the patient had no mucositis. A follow-up evaluation was performed a month after discharge the patient. Unusual clinical presentation was addressed whenever observed.

Criteria for evaluation:

Primary efficacy variable:

o Rate of absent of mucositis at any of the visits using WHO scale for mucositis and OMAS.

Secondary efficacy variables:

* Severity of oral mucositis at any of the visits using WHO scale for mucositis and OMAS.
* Severity of oral pain at any of the visits using WHO scale for mucositis and OMAS.
* Safety (oral adverse events)
* Patients' acceptance of the study drug on an 11-step ladder. Others
* Compliance with standard oral care (chlorhexidine rinse, nystatin readymix, saline mouthwash)

ELIGIBILITY:
Inclusion Criteria:

* No oral ulceration at baseline
* At risk for oral mucositis due to the conditioning regimen to HSCT
* Age above 18 years old
* Karnofsky score >60
* Agree to participate in the study (signed an informed consent)

Exclusion Criteria:

* Pregnant woman
* Well-founded doubt about the patient's jurisprudence
* Children
* Sensitivity to light or treated with drugs which are sensitizers to light
* Treatment with other experimental topical drug during the study period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual)